CLINICAL TRIAL: NCT03728374
Title: Anlotinib Hydrochloride as Second-line Therapy in Elderly Patients With EGFR Wild-type Lung Adenocarcinoma Who Refused Chemotherapy: an Open, Single-arm, Single-center Clinical Trial
Brief Title: Anlotinib Hydrochloride as Second-line Therapy in Elderly Patients With EGFR Wild-type Lung Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Hanyan Xu, professor, First Affiliated Hospital of Wenzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FirstWenzhouMU
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Non-Small-Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib (Experimental)
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — Anlotinib ( 12mg, QD, PO, d1-14, 21 days per cycle)

SUMMARY:
Anlotinib is a multi-target receptor tyrosine kinase inhibitor in domestic research and development. It can inhibit the angiogenesis related kinase, such as VEGFR, FGFR, PDGFR, and tumor cell proliferation related kinase -c-Kit kinase. In the phase Ⅲ study, patients who failed at least two kinds of systemic chemotherapy (third line or beyond) or drug intolerance were treated with anlotinib（12mg，po. qd. on day 1to14 of a 21-day cycle） or placebo, the anlotinib group PFS and OS were 5.37 months and 9.63 months, the placebo group PFS and OS were 1.4 months and 6.3 months. Subgroup analysis results suggest that elderly patients may get longer mPFS and mOS.

Therefore, the investigators envisage an open, single-arm, single-center clinical trial using anlotinib in elderly patients with EGFR wild-type lung adenocarcinoma who refused chemotherapy, to find if anlotinib is a better option in NSCLC second-line therapy.

DETAILED DESCRIPTION:
It is an open, single-arm, single-center clinical trial conducted in China, and plan to Recruiting 38 patients (≥65 years old, ECOG PS 0-2) who were progressed after first line systemic therapy and refused/can't tolerate chemotherapy. Patents receive 12mg anlotinib orally daily on day 1to 14 of a 21-day cycle until progression of disease, assess safety and efficacy of the drug.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects voluntarily joined the study and signed informed consent, with good compliance and follow-up;
* 2. Diagnosed as locally advanced and / or metastatic non-small cell lung adenocarcinoma (NSCLC) by cytology or histology; diagnosed as stage IIIB, IIIC or IV according to the 2017 new version of the UICC lung cancer staging criteria (8th edition); : Patients with stage IIIB and IIIC must be at least one measurable lesion in patients who cannot be surgically resected according to RECIST 1.1;
* 3. For local advanced or metastatic NSCLC, disease progression occurred after first-line systemic treatment previously;
* 4. Provide detectable specimens (tissue or cancerous pleural effusion) for genotyping before enrollment, and the patients should be with negative EGFR, ALK, and ROS1 gene test results;
* 5. The patient refuses to receive second-line chemotherapy (such as docetaxel, pemetrexed, etc.); or is assessed to be unable to tolerate second-line chemotherapy;
* 6. Age ≥ 65 years old, ECOG PS 0-2 points;
* 7. At least one target lesion that has not received radiotherapy in the past 3 months, and accurate measurement by magnetic resonance imaging (MRI) or computed tomography (CT) in at least 1 direction (maximum diameter required to be recorded) (conventional CT ≥ 20 mm or ≥ 10 mm under spiral CT);
* 8. Life expectancy is at least 3 months;
* 9. The damage subjects received from other treatments has recovered(NCI-CTCAE version 4.0 grade ≤ 1), the interval of subjects receiving nitrosourea or mitomycin should be at least 6 weeks; the interval subjects receiving other cytotoxic drugs, bevacate Avastin (Avastin), surgery should be at least 4 weeks; the interval subjects receiving radiotherapy (except for local palliative radiotherapy) should be at least 2 weeks;
* 10. The main organs function are normally, the following criteria are met: (1) Blood routine examination criteria should be met (no blood transfusion and blood products within 14 days, no correction by G-CSF and other hematopoietic stimuli): HB≥90 g/L; ANC ≥ 1.5×10^9/L; PLT ≥80×10^9/L; (2) Biochemical examinations must meet the following criteria: TBIL<1.5×ULN; ALT and AST < 2.5×ULN, and for patients with liver metastases < 5×ULN; Serum Cr ≤ 1.25×ULN or endogenous creatinine clearance > 60 ml/min (Cockcroft-Gault formula).

Exclusion Criteria:

* 1. Small cell lung cancer (including lung cancer mixed with small cell lung cancer and non-small cell lung cancer);
* 2. Lung squamous cell carcinoma, or non-small cell lung cancer with hemoptysis (>50 ml / day);
* 3. Imaging (CT or MRI) shows that the distance between tumor lesion and the large blood vessel is ≤ 5 mm, or there is a central tumor that invades the local large blood vessel; or there is a significant pulmonary cavity or necrotizing tumor;
* 4. Elderly patients who have been evaluated to be able to tolerate second-line chemotherapy
* 5. Allergic reactions to allosterinib or excipients in the test drug;
* 6. A patient who develops an allergic reaction to contrast agent;
* 7. History and comorbidities

  1) Active brain metastases, cancerous meningitis, spinal cord compression, or imaging CT or MRI screening for brain or pia mater disease (a patient with brain metastases who have completed treatment and stable symptoms in 28 days before enrollment may be enrolled, but should be confirmed by brain MRI, CT or venography evaluation as no cerebral hemorrhage symptoms); 2) The patient is participating in other clinical studies or completing the previous clinical study in less than 4 weeks; 3) Other active malignancies that require simultaneous treatment; 4) Patients with a history of malignant tumors except for patients with cutaneous basal cell carcinoma, superficial bladder cancer, cutaneous squamous cell carcinoma or orthotopic cervical cancer who have undergone a curative treatment and have no disease recurrence within 5 years from the start of treatment 5) Patients with previous anti-tumor treatment-related adverse reactions (excluding hair loss) who have not recovered to NCI-CTCAE ≤1; 6) Abnormal blood coagulation (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or APTT > 1.5 ULN), with bleeding tendency or undergoing thrombolytic or anticoagulant therapy; 7) Note: Under the premise of prothrombin time international normalized ratio (INR) ≤ 1.5, low-dose heparin (adult daily dose of 0.6 million to 12,000 U) or low-dose aspirin (daily dosage ≤ 100 mg) is allowed for preventive purposes; 8) Renal insufficiency: urine routine indicates urinary protein ≥ ++, or confirmed 24-hour urine protein ≥ 1.0g; 9) Uncontrollable hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg, despite optimal medical treatment); 10) The effects of surgery or trauma have been eliminated for less than 14 days before enrollment in subjects who have undergone major surgery or have severe trauma; 11) Severe acute or chronic infections requiring systemic treatment; 12) Suffering from severe cardiovascular disease: myocardial ischemia or myocardial infarction above grade II, poorly controlled arrhythmias (including men with QTc interval ≥ 450 ms, women ≥ 470 ms); according to NYHA criteria, grades III to IV Insufficient function, or cardiac color Doppler ultrasound examination indicates left ventricular ejection fraction (LVEF) <50%; 13) There is currently a peripheral neuropathy of ≥CTCAE 2 degrees, except for trauma; 14) Respiratory syndrome (≥CTC AE grade 2 dyspnea), serous effusion (including pleural effusion, ascites, pericardial effusion) requiring surgical treatment; 15) Long-term unhealed wounds or fractures; 16) Severe weight loss (greater than 10%) within 6 weeks prior to randomization; 17) Decompensated diabetes or other ailments treated with high doses of glucocorticoids; 18) Factors that have a significant impact on oral drug absorption, such as inability to swallow, chronic diarrhea, and intestinal obstruction; 19) Clinically significant hemoptysis (daily hemoptysis greater than 50ml) within 3 months prior to enrollment; or significant clinically significant bleeding symptoms or defined bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood ++ and above, or suffering from vasculitis; 20) Events of venous/venous thrombosis occurring within the first 12 months prior to enrollment, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism; 21) Planned for systemic anti-tumor therapy, including cytotoxic therapy, signal transduction inhibitors, immunotherapy (4 weeks prior to enrollment in other anti-cancer drug clinical trials or within 4 weeks prior to grouping or during the study period Or use mitomycin C) within 6 weeks prior to receiving the test drug. Radiation-rehabilitation radiotherapy (EF-RT) was performed within 4 weeks before grouping or limited-field radiotherapy to be evaluated for tumor lesions within 2 weeks before grouping.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
PFS | each 42 days up to PD or death(up to 24 months)
  Progress free survival

SECONDARY OUTCOMES:
OS | From randomization until death (up to 24 months)
  Overall Survival
ORR | Time Frame: each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Objective Response Rate
DCR | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Disease Control Rate
QoL: EORTC QLQ-C30 | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  use EORTC QLQ-C30(version 3) questionnaire to evaluate the quality of life
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Until 21 day safety follow-up visit
  Record Adverse Events (AEs) according to CTCAE (V4.03). To find Potential adverse reaction, measure blood pressure at least 2 times a week and test blood routine, Blood biochemical, Urine routine, stool routine, coagulation function, electrocardiogram for each follow-up, record and analyze the number of abnormal data.

CONTACTS AND LOCATIONS:
Overall Officials: Yuping Li, doctor, Study Chair — First Affiliated Hospital of Wenzhou Medical University

IPD SHARING:
Plan to Share IPD: No